CLINICAL TRIAL: NCT06930209
Title: Histological Analysis of CelluJuve® Injected Into the Brachium of Healthy Volunteers
Brief Title: Histological Analysis of CelluJuve® Injections in the Brachium
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spiderwort Biotechnologies Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPDR-2023-002
Record Dates: First submitted 2025-03-21; First posted 2025-04-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Male and Female Subjects
Keywords: Histological Analysis; Dermal Filler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CelluJuve® (Experimental)
  Interventions: Device: CelluJuve®

INTERVENTIONS:
Device: CelluJuve® — CelluJuve® injected into upper brachium

SUMMARY:
Single-center, exploratory study assessing the safety and histological presentation of CelluJuve® injected into the brachium of healthy volunteers

DETAILED DESCRIPTION:
At Visit 1 (Baseline), all subjects will receive injections (0.2mL bolus) of CelluJuve® into the proximal medial aspect of the brachium of their non dominant arm. The volume per microbolus of CelluJuve® into a single injection site is 0.2 mL. All injections will be performed using the same type/brand of 25G x 1/2" (0.50x13 mm) needle.

One 5-mm punch biopsy will be taken from injection sites at 2 weeks, 1 month and 3 months. Punch biopsy samples will be fixed in formol before being frozen or dehydrated, impregnated in paraffin, and embedded. Prepared samples will then be cut into 4 µm sections and analyzed for general morphology, immunostaining, and immunogenicity. Analysis will be performed at the epidermis, papillary dermis, and lower reticular dermis depending on the extracellular matrix component of interest.

Safety will be assessed through AE reporting, study diaries, and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers of any race between 30 and 65 years of age.
2. Female subjects of childbearing potential must have a negative UPT at Visit 1 and practice a reliable method of contraception throughout the study.
3. Healthy skin in the study treatment area and free of conditions or diseases that could interfere with study evaluations.
4. Subjects willing to receive microbolus injections of CelluJuve® into the proximal medial aspect of the brachium of their non-dominant arm, and willing to have one 5-mm cutaneous punch biopsy taken from each injection site.
5. Able to follow study instructions and complete all required visits.
6. Signed ICF and Photographic Release.

Exclusion Criteria:

1. Female subjects that are pregnant, breast-feeding, or of childbearing potential and not practicing reliable contraception.
2. Study staff or close relative to study staff (e.g., parents, children, siblings, or spouse).
3. Subjects with known prolonged bleeding times due to disease or ongoing regimen use of anticoagulants (e.g., warfarin).
4. Acute or chronic skin disease, inflammation, or related conditions, cancerous or precancerous lesions near the treatment area.
5. Presence of any skin pathology or condition that could interfere with the evaluation of the treatment areas, worsen due to study treatment, or require interfering topical, systemic, or surgical therapy.
6. Known history of medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with interpretation of study results or compliance of the subject and could make the subject inappropriate for study entry.
7. Known history of allergic/anaphylactic reactions to any of the components of CelluJuve® including known sensitivity to cellulose, porcine gelatin, or to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
8. Known history of malignancy (excluding non-melanoma skin cancer) within the past 3 years.
9. Known history of systemic granulomatous diseases active or inactive (e.g., Sarcoid, Wegener's disease, TB, etc.) or connective tissue diseases (e.g., lupus, dermatomyositis, etc.).
10. Known history or evidence of keloid scarring, susceptibility to keloid formation or hypertrophic scarring, or delayed healing activity.
11. Known history or presence of severe chronic systemic diseases, including but not limited to, poorly controlled diabetes mellitus (all types), congestive heart failure, severe liver disease, severe kidney disease, and others as judged by the Investigator.
12. Known history or presence of any autoimmune or connective tissue disease, receiving treatment with immunomodulating therapy, or is immunocompromised or immunosuppressed.
13. Known history of clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
14. Undergoing, or planning to undergo, radiation or ultrasound therapy in the treatment area.
15. Unwilling to adhere to medication restrictions for the duration of the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Histological assessment of biopsies - general morphology | 3 months
  Assessment of general morphology (e.g., Masson's trichrome)
Histological assessment of biopsies - immunostaining | 3 months
  Assessment of immunostaining (e.g., collagen, elastin, etc.)
Histological assessment of biopsies - immunogenicity | 3 months
  Assessment of immunogenicity (e.g., inflammatory markers, cytokines, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- BioPharma Services Inc., North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No